CLINICAL TRIAL: NCT07081698
Title: Walnut as a First Food During Complementary Feeding on Gut Microbiota and Immunity Development in Breastfed Infants
Brief Title: Walnuts as an Infant Solid Food for Health
Acronym: WISH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado State University (Other)
Collaborators: California Walnut Commission (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Basic Science
Other Study IDs: 6690
Record Dates: First submitted 2025-02-27; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Gut -Microbiota; Inflammatory Markers; Infant Development
Keywords: Walnut; Microbiome; Infant; Pediatric; Nutrition; Health

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The walnut group (Experimental): The intervention group will provide 10g of walnuts daily to their infant for 7 months.
  Interventions: Other: Infant walnut intake
- Control Group (No Intervention): The control group will be asked to limit walnuts and tree nuts.

INTERVENTIONS:
Other: Infant walnut intake — The intervention group will receive walnuts at 10 g/day, and the control group will be advised to avoid walnuts/tree nuts during the intervention. The purpose of this research is to learn more about how walnuts as a first food in infants impact immunity and the development of bacteria living in your baby's gut.
  Arms: The walnut group

SUMMARY:
The objective is to investigate the effect of walnuts on gut microbiota, inflammatory markers, atopic dermatitis status, and indices of allergy outcomes in breastfed infants during early complementary feeding.

The three primary aims include:

Aim 1: Evaluate the effect of walnut consumption on gut microbiota structure and function, inflammation, atopic dermatitis, and allergy outcomes.

Aim 2: Evaluate the impact of walnut consumption on infant growth trajectories and risk of overweight.

Aim 3 (exploratory): Identify walnut-specific food signatures that are associated with gut microbiota and immunity biomarkers using a novel nutri-metabolomics technique.

DETAILED DESCRIPTION:
Some details are intentionally left to out to preserve the scientific integrity of the study, and they will be included in the record after the study is completed.

ELIGIBILITY:
Inclusion Criteria:

* Full term: gestational age ≥ 37 weeks
* Generally healthy without conditions that would affect normal growth
* No significant consumption of complementary food (e.g., no more than 1 oz of solid foods per week)
* Exclusively breastfed (< 2 weeks of cumulative formula exposure)

Exclusion Criteria:

* Adults unable to consent
* Pregnant women
* Prisoners

Ages: 5 Months to 5 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2025-05-18 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Gut Microbiome Composition Analyzed using 16S rRNA Amplicon Sequencing | Over 7 months
  16S rRNA amplicon sequencing is used to profile taxonomic makeup of fecal specimens. Within the gut microbiome composition, microbial diversity will be summarized using common ecological measures (Good's coverage, Sobs, and Shannon alpha diversity).
Infant Growth (Length) | Over 7 months
  Measured in cm
Infant Growth (Weight) | Over 7 months
  Measured in kg
Dietary Intake | Over 7 months
  3 day dietary recall with results generated by NDSR software
IL-33 (Interleukin-33) | Over 7 months
  Measured in pg/mL
IL-6 (Interleukin-6) | Over 7 months
  Measure in pg/mL
IL-8 (Interleukin-8) | Over 7 months
  Measured in pg/mL
IL-13 (Interleukin-13) | Over 7 months
  Measured in pg/mL
TGF-b (Transforming growth factor beta) | Over 7 months
  Measured in ng/ml.
IL-4 (Interleukin-4) | Over 7 months
  Measured in pg/mL
IL-10 (Interleukin 10) | Over 7 months
  Measured in pg/mL

SECONDARY OUTCOMES:
Walnut-Specific Food Signatures (Compounds) as Assessed by Metabolomics Analysis | Over 7 months
  Metabolomics analysis (nutri-metabolomics) is used to identify and validate food-derived biomarkers that may be classified as biomarkers of intake and/or biomarkers of effect, both of which can be linked to health indicators.

CONTACTS AND LOCATIONS:
Overall Officials: Minghua Tang, Phd, Principal Investigator — Colorado State University
Locations (1):
- Food Science and Human Nutrition Clinical Research Laboratory, Fort Collins, Colorado, United States

IPD SHARING:
Plan to Share IPD: No